CLINICAL TRIAL: NCT05563870
Title: A Combined Endoscopy and Radiology-guided Radiofrequency Ablation Therapy Protocol for Inoperable Perihilar Cholangiocarcinoma
Brief Title: Endoscopy and Radiology-guided Ablation for Inoperable Cholangiocarcinoma
Acronym: COMBO-RFA
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Clinical Hospital Colentina (Other)
Collaborators: Carol Davila University of Medicine and Pharmacy (Other); Universitatea din Bucuresti (Other)
Responsible Party: Principal Investigator, dr. Theodor Alexandru Voiosu, Gastroenterology Consultant, Clinical Hospital Colentina
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: COMBO-RFA
Record Dates: First submitted 2022-09-20; First posted 2022-10-03 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2024-03

CONDITIONS: Perihilar Cholangiocarcinoma
Keywords: perihilar cholangiocarcinoma; ERCP; Radiofrequency ablation
MeSH Terms: conditions — Klatskin Tumor

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Endoscopic Drainage Arm (Active Comparator): Patients randomized to this arm will undergo biliary stenting only
  Interventions: Procedure: Endoscopic biliary stenting
- COMBO-RFA Arm (Experimental): Patients randomized to this arm will undergo same-session endoluminal radiofrequency ablation followed by biliary stenting
  Interventions: Procedure: Endoluminal radiofrequency ablation; Procedure: Endoscopic biliary stenting

INTERVENTIONS:
Procedure: Endoluminal radiofrequency ablation — Endoluminal Radiofrequency ablation (RFA) of the entire stricture length will be performed using the Habib probe. A current of 7W will be delivered for 90s intervals at a time. If multiple ablation sessions are needed in order to ablate the entire stricture lenght, there will be an overlap of ablated areas in order to ensure proper stricture treatment. Dilation of the stricture prior to RFA delivery will be performed if required. After RFA treatment, biliary drainage of all hepatic territories will be ensured.
  Arms: COMBO-RFA Arm
Procedure: Endoscopic biliary stenting — Endoscopic biliary stenting will be performed via ERCP using multiple plastic stents, in order to ensure propper drainage of all accessed hepatic territories.

SUMMARY:
This prospective clinical trial aims to assess the feasibility, efficacy, and safety of a personalized radiofrequency ablation protocol coupled with complete biliary drainage for patients presenting with inoperable perihilar cholangiocarcinoma.

DETAILED DESCRIPTION:
This clinical trial proposes a personalized treatment approach to inoperable perihilar cholangiocarcinoma consisting of endoluminal ablative therapy via radiofrequency ablation followed by endoscopic biliary drainage.

Patients presenting with jaundice / biliary obstruction caused by inoperable perihilar cholangiocarcinoma as assessed during multidisciplinary case discussion will be invited to enroll in this trial.

Patients will be randomized in a 1:1 fashion to receive biliary plastic stenting (control arm) or biliary plastic stenting + radiofrequency ablation via endoscopic approach. In cases where ERCP fails to achieve adequate biliary drainage, stenting and/or drainage will be attempted via percutaneous approach.

Additional systemic chemotherapy will be offered to all eligible patients according to the local standard of care.

Patients will be followed up with a clinical visit at 2 weeks and stent exchange (+ additional RFA treatment in the control arm) will be offered at 8-12 weeks interval until disease progression, clinical deterioration precluding ERCP or death.

The main study objectives are:

* To assess the technical feasibility of implementing the proposed therapeutic protocol involving a combined endoscopic-radiologic approach to drainage and ablation
* To evaluate the efficacy of radiofrequency ablation in local disease control
* To evaluate whether complete drainage and radiofrequency ablation have a cumulative benefit in patients with inoperable perihilar cholangiocarcinoma
* To evaluate the safety of our proposed therapeutic protocol combining interventional endoscopy with radiology

ELIGIBILITY:
Inclusion Criteria:

* perihilar cholangiocarcinoma
* locally advanced disease (unresectable)
* M1 (limted to 1 site)

Exclusion Criteria:

* refusal to sogn the ICF
* poor performance status (ECOG >2)
* surgically altered anatomy (i.e Bilroth II or Roux-en-Y interventions)
* significant comorbidities
* ASA score >3
* life expectancy <3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2024-10-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Technical success of ERCP procedure | 2 months
  Ability to correctly apply radiofrequency ablation and place stents in all the biliary ducts accessed on ERCP
Tumor response | 6 months
  To evaluate the efficacy of radiofrequency ablation in local disease control by assessing tumor response according to RECIST criteria at 6 months follow-up

SECONDARY OUTCOMES:
Rate of procedure-related adverse events | 12 months
  To evaluate the safety profile of the procedure by assessing the rate of procedure-related adverse events according to the ASGE lexicon (cholangitis, bleeding, perforation, pancreatitis) after endoscopic treatment
Overall survival | 12 months
  To assess patient survival rates at 12 months follow-up
Tumor microenvironment alterations | 2 months
  To evaluate the expression of programmed death (PD)-1 / PD- ligand 1 markers on biopsy samples of tumor tissue obtained at the index and follow-up ERCP procedure

CONTACTS AND LOCATIONS:
Locations (1):
- Gastroenterology Department, Colentina Hospital, Bucharest, Romania

IPD SHARING:
Plan to Share IPD: No